CLINICAL TRIAL: NCT06270810
Title: Cardiometabolic Effects of Increasing Non-Exercise Physical Activity Combined With Aerobic Exercise in Overweight Young Women
Brief Title: Cardiometabolic Effects of Combined Aerobic Exercise and Non-Exercise Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Yasin Ak, Principal Investigator, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Aero-PA
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Overweight
Keywords: Overweight; non-Exercise Physical Activity; Aerobic Exercise; Sedentary Behaviour; Physical Activity; Step Counts; Cardiometabolic; Blood Lipids; Serum Glucose; HbA1c; Blood Pressure; Young Women; Cardiorespiratory Fitness
MeSH Terms: conditions — Overweight; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise (AeroEx) Group (Experimental): Participants in this group will do moderate-intensity aerobic training for 4 days a week for 8 weeks.
  Interventions: Behavioral: Aerobic Exercise
- Aerobic Exercise+non-Exercise (nE) Physical Activity (AeroEx+nE PA) Group (Experimental): Participants in this group will increase their non-exercise physical activities and do moderate-intensity aerobic training for four days a week for 8 weeks.
  Interventions: Behavioral: Aerobic Exercise; Behavioral: Increasing non-Exercise Physical Activity

INTERVENTIONS:
Behavioral: Aerobic Exercise — Aerobic exercise will be performed on the treadmill at 40-60% of the participants' heart rate reserves. Each aerobic exercise session will last for 40 minutes. All participants will be monitored with a heart rate monitor throughout the exercise sessions. During the first three-week, participants will exercise on the treadmill at intensities between 40-50%, and between fourth and eighth weeks, 50-60% of their heart rate reserves. Participants will wear an accelerometer on their non-dominant wrist during the intervention to monitor the physical activity and sedentary behavior data. At the same time, these participants will be asked not to change their routine diet during the intervention period.
Behavioral: Increasing non-Exercise Physical Activity — Participants who will carry out this intervention will increase their non-exercise physical activities. Before intervention period, participants will receive face-to-face training to increase their non-exercise physical activities. This training will generally consist of recommendations based on the study which effectively reduced sedentary behavior (SB) with non-exercise physical activities (Sarah Kozey-Keadle et al. 2012). A one-on-one interview will be held with each participant every week to learn about strategies by which the volunteers successfully increased their non-exercise physical activities in the previous week, and the difficulties or barriers they encountered. New strategies to overcome these difficulties and barriers will be discussed and suggestions will be made. Participants will wear an accelerometer on their non-dominant wrist to monitor the physical activity and SB data, and will be asked not to change their routine diet during the intervention period.
  Arms: Aerobic Exercise+non-Exercise (nE) Physical Activity (AeroEx+nE PA) Group

SUMMARY:
The goal of this clinical trial is to investigate whether increasing non-exercise physical activity combined with aerobic exercise in overweight young women is superior to performing aerobic exercise alone in terms of some cardiometabolic variables.

The main question it aims to answer is:

• Do both increasing non-exercise physical activity and doing aerobic exercise add more beneficial cardiometabolic effects to performing aerobic exercise alone in overweight young women?

To answer this question, overweight young women will be randomly assigned to two different groups of this research. Volunteers in one of the groups will do moderate-intensity aerobic training and the other group will increase their non-exercise physical activities in addition to moderate-intensity aerobic training. Then researchers will compare two groups to see the differences in cardiometabolic variables.

DETAILED DESCRIPTION:
According to objective and subjective measurements, time spent sedentary varies between 2.5 hours and 10 hours approximately in European countries. In America, this time is 8.44 hours on average. According to accelerometer data, the average total sedentary time of university students is 9.82 hours per day. Sedentary behaviour (SB) is associated with cardiometabolic risk markers and increased risk of cardiovascular disease, independent of moderate and vigorous physical activity (PA). Replacing sedentary time with PA of any intensity, including low-intensity, reduces all-cause mortality.

In terms of some cardiovascular risk variables (e.g., high triglycerides, glucose, LDL cholesterol, total cholesterol), data are insufficient and conflicting on the superiority of increasing non-exercise PA in addition to aerobic exercise over aerobic exercise alone. Additionally, to our knowledge, whether increasing non-exercise PA combined with aerobic exercise is superior to performing aerobic exercise alone in young overweight women with high sedentary time has not been investigated. Therefore, this study was planned to investigate whether reducing SB and increasing non-exercise PA combined with aerobic exercise in overweight young women between the ages of 18-35 is superior to performing aerobic exercise alone in terms of some cardiometabolic variables. For this purpose, overweight female individuals between the ages of 18-35 will be invited to the research. Thirty-two female volunteers who meet the inclusion and exclusion criteria will be randomly assigned to two different groups of this research. These groups will be as follows:

Aerobic Exercise Group: Participants in this group will do moderate-intensity aerobic training four days a week for 8 weeks.

Aerobic Exercise+non-Exercise Physical Activity Group: Participants in this group will reduce their sedentary time and increase non-exercise PA in addition to moderate-intensity aerobic training for four days a week for 8 weeks.

PA and SB data of the participants in both groups will be monitored with a wrist worn accelerometer throughout the study. At the beginning of the study, 4 weeks after the beginning and at the end of 8 weeks, participants will be evaluated in terms of the cardiometabolic variables. These variables are fasting serum glucose, triglyceride, HDL cholesterol, LDL cholesterol, HbA1c, systolic blood pressure, diastolic blood pressure, cardiorespiratory fitness, body mass index, waist and hip circumference, and body fat percentage. If there is a difference between the two group averages in terms of all variables and the group-time interactions test assumptions are met, analysis will be made with two-way mixed analysis of variance (ANOVA). Since 3 measurements will be made over time, pairwise differences in change over time will be analyzed with a post hoc Bonferroni test.

ELIGIBILITY:
Inclusion Criteria:

* To have a body mass index between 25 kg.(m2)-1 and 29.9 kg.(m2)-1
* Self reported sitting time greater than 7 hours per day
* Not exercising regularly in the last 3 months

Exclusion Criteria:

* Hypertension
* Coronary heart disease
* Heart failure
* Diabetes mellitus (A1C being 6.5% and above)
* Prediabetes (A1C between 5.7% and 6.4%)
* Metabolic syndrome
* Hypothyroidism
* Non-alcoholic fatty liver disease
* Chronic inflammatory disease
* Chronic renal failure
* Cushing's syndrome
* Musculoskeletal disorder that will affect the ability to do physical activity
* HIV infection
* Being on antihypertensive medication
* Being on lipid-lowering medication
* Being on antidiabetic medication
* Being on systemic glucocorticoid medication
* Smoking
* Pregnancy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Low Density Lipoprotein (LDL) Cholesterol | The week before the beginning of the interventions, at 4th week of the intervention , and the week after the interventions
  Fasting blood samples will be taken by applying a vacutainer needle to the appropriate vein following a 12-hour fast and will be analyzed immediately in the biochemistry laboratory.
High Density Lipoprotein (HDL) Cholesterol | The week before the beginning of the interventions, at 4th week of the intervention , and the week after the interventions
  Fasting blood samples will be taken by applying a vacutainer needle to the appropriate vein following a 12-hour fast and will be analyzed immediately in the biochemistry laboratory.
Total Cholesterol | The week before the beginning of the interventions, at 4th week of the intervention , and the week after the interventions
  Fasting blood samples will be taken by applying a vacutainer needle to the appropriate vein following a 12-hour fast and will be analyzed immediately in the biochemistry laboratory.
Glycated Hemoglobin (HbA1C) | The week before the beginning of the interventions, at 4th week of the intervention , and the week after the interventions
  Fasting blood samples will be taken by applying a vacutainer needle to the appropriate vein following a 12-hour fast and will be analyzed immediately in the biochemistry laboratory.
Serum Triglycerides | The week before the beginning of the interventions, at 4th week of the intervention , and the week after the interventions
  Fasting blood samples will be taken by applying a vacutainer needle to the appropriate vein following a 12-hour fast and will be analyzed immediately in the biochemistry laboratory.
Maximal Oxygen Consumption | The week before the beginning of the interventions, and the week after the interventions
  Maximal oxygen consumption will be estimated by the Rockport 1 Mile Walk Test
Systolic Blood Pressure | The week before the beginning of the interventions, at 4th week of the intervention , and the week after the interventions
  Measurements will be made on the arm with a digital blood pressure monitor after resting for at least 10 minutes in a supine position to ensure hemodynamic stability. By wrapping the cuff around the arm, brachial systolic blood pressure will be automatically measured.
Diastolic Blood Pressure | The week before the beginning of the interventions, at 4th week of the intervention , and the week after the interventions
  Measurements will be made on the arm with a digital blood pressure monitor after resting for at least 10 minutes in a supine position to ensure hemodynamic stability. By wrapping the cuff around the arm, brachial diastolic blood pressure will be automatically measured.

SECONDARY OUTCOMES:
Body Fat Percentage | The week before the beginning of the interventions, at 4th week of the intervention , and the week after the interventions
  Body fat percentage will be measured by bioelectrical impedance analysis
Fat-free Mass | The week before the beginning of the interventions, at 4th week of the intervention , and the week after the interventions
  Fat-free mass will be measured by bioelectrical impedance analysis
Waist Circumference | The week before the beginning of the interventions, at 4th week of the intervention , and the week after the interventions
  Waist circumference will be measured in centimeters in the horizontal plane with a tape measure from the narrowest part of the waist area, with feet together, immediately after normal expiration without holding the breath.
Hip Circumference | The week before the beginning of the interventions, at 4th week of the intervention , and the week after the interventions
  Hip circumference will be measured in centimeters in the horizontal plane with a tape measure from the widest part of the hip.

CONTACTS AND LOCATIONS:
Locations (1):
- Kastamonu University, Çatalzeytin Vocational School, Çatalzeytin, Kastamonu, Turkey (Türkiye)

REFERENCES:
- [Background] Kozey-Keadle S, Libertine A, Staudenmayer J, Freedson P. The Feasibility of Reducing and Measuring Sedentary Time among Overweight, Non-Exercising Office Workers. J Obes. 2012;2012:282303. doi: 10.1155/2012/282303. Epub 2011 Nov 16. PMID 22175004
- [Background] Kozey Keadle S, Lyden K, Staudenmayer J, Hickey A, Viskochil R, Braun B, Freedson PS. The independent and combined effects of exercise training and reducing sedentary behavior on cardiometabolic risk factors. Appl Physiol Nutr Metab. 2014 Jul;39(7):770-80. doi: 10.1139/apnm-2013-0379. Epub 2014 Jan 7. PMID 24971677